CLINICAL TRIAL: NCT04580628
Title: Thuflep/SOLEP : Initial Experience and Results of Prostate Laser Enucleation With Thulium-fiber Laser (TFL)
Status: Completed | Type: Observational
Sponsor: Clinique Saint-Hilaire (Other)
Responsible Party: Principal Investigator, MALVAL Benoit, Principal Investigator, Doctor in urology department, Clinique Saint-Hilaire
Other Study IDs: 202000549
Record Dates: First submitted 2020-09-19; First posted 2020-10-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thuflep TLF: initial experience and results of prostate laser enucleation with fibrous thulium laser (TLF)

DETAILED DESCRIPTION:
While prostate laser enucleation is being confirmed as the new gold standard for surgical management of benign prostate hypertrophy, the holmium:Yag laser is currently the most widely used. A new laser technology, the fibrous thulium laser (TFL), has recently appeared with clearly superior results for lithotripsy. The question therefore arises of the surgical and functional results of the use of fibrous thulium for prostate enucleation.

ELIGIBILITY:
Inclusion Criteria:

* Patients superior or equal to 18 years old
* Benign Prostate Hypertrophy ( more than 30cc.)
* Indication to surgical treatment
* No contraindication for surgery
* No opposition to participating in the study

Exclusion Criteria:

* Evidence of urethral stenosis
* Evidence of a bladder tumour
* Evidence of prostate cancer known or confirmed by prostate biopsies if suspected
* Known neurological bladder
* Refusal to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients treated at clinique saint hilaire Rouen with Thuflep, who consent
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring the evolution of Urinary Symptoms Rated by the IPSS Score after prostate laser enucleation with TFL | MONTH 12
  self reported International Prostate Symptom Score (IPSS) From 0 (no symptom) to 35 (maximum symptoms)

SECONDARY OUTCOMES:
Rate of post-operative complications | MONTH 6
  post operative complications : urethral stenosis, prostate bed sclerosis, overactive bladder, urinary incontinence, erectile dysfunction
duration of intervention | POST SURGERY HOUR 24
  in minutes
bloodloss assessment | Day 1
  measurement of haemoglobinemia
max flow assessment | MONTH 12
  measured with urinary flowmeter in ml/sec
max flow assessment | MONTH 6
  measured with urinary flowmeter
max flow assessment | MONTH 3
  measured with urinary flowmeter
max flow assessment | MONTH 1
  measured with urinary flowmeter
post-void residual (PVR) urine test | MONTH 12
  ml
post-void residual (PVR) urine test | MONTH 6
  ml
post-void residual (PVR) urine test | MONTH 3
  ml
post-void residual (PVR) urine test | MONTH 1
  ml
erectile dysfunction assessment | MONTH 12
  self reported International Index of Erectile Function 5 score(IIEF-5) from 5 : severe erectil dysfunction to 25 : no erectile dysfunction
erectile dysfunction assessment | MONTH 6
  self reported International Index of Erectile Function 5 score(IIEF-5) from 5 : severe erectil dysfunction to 25 : no erectile dysfunction
erectile dysfunction assessment | MONTH 3
  self reported International Index of Erectile Function 5 score(IIEF-5) from 5 : severe erectil dysfunction to 25 : no erectile dysfunction
erectile dysfunction assessment | MONTH 1
  self reported International Index of Erectile Function 5 score(IIEF-5) from 5 : severe erectil dysfunction to 25 : no erectile dysfunction
quality of life assessment | MONTH 12
  self reported Short Form (36) Health Survey score(SF-36) from 0 to 100 (good health)
quality of life assessment | MONTH 6
  self reported Short Form (36) Health Survey score(SF-36) from 0 to 100 (good health)
quality of life assessment | MONTH 3
  self reported Short Form (36) Health Survey score(SF-36) from 0 to 100 (good health)
quality of life assessment | MONTH 1
  self reported Short Form (36) Health Survey score(SF-36) from 0 to 100 (good health)
urinary incontinence Assessment | MONTH 12
  self reported International Consultation on Incontinence: short questionary score (ICIQ) from 0 : no leaks, to 19 : major leaks
urinary incontinence Assessment | MONTH 6
  self reported International Consultation on Incontinence: short questionary score (ICIQ) from 0 : no leaks, to 19 : major leaks
urinary incontinence Assessment | MONTH 3
  self reported International Consultation on Incontinence: short questionary score (ICIQ) from 0 : no leaks, to 19 : major leaks
urinary incontinence Assessment | MONTH 1
  self reported International Consultation on Incontinence: short questionary score (ICIQ) from 0 : no leaks, to 19 : major leaks
prostatic specific antigen in ng/mL level evolution | MONTH 1
  ng/ml
Measuring the evolution of Urinary Symptoms Rated by the IPSS Score after prostate laser enucleation with TFL | MONTH 1
  self reported International Prostate Symptom Score (IPSS) From 0 (no symptom) to 35 (maximum symptoms)
Measuring the evolution of Urinary Symptoms Rated by the IPSS Score after prostate laser enucleation with TFL | MONTH 3
  self reported International Prostate Symptom Score (IPSS) From 0 (no symptom) to 35 (maximum symptoms)
Measuring the evolution of Urinary Symptoms Rated by the IPSS Score after prostate laser enucleation with TFL | MONTH 6
  self reported International Prostate Symptom Score (IPSS) From 0 (no symptom) to 35 (maximum symptoms)
PATIENT GLOBAL IMPRESSION OF IMPROVEMENT | MONTH 1
  SELF REPORT SATISFACTION QUESTIONARY FROM 1 (better condition ) to 7 ( worse condition)
PATIENT GLOBAL IMPRESSION OF SEVERITY | MONTH 1
  SELF REPORT SATISFACTION QUESTIONARY FROM 1( normal )to 4 (severe )

CONTACTS AND LOCATIONS:
Overall Officials: BENOIT MALVAL, Principal Investigator — Clinique Saint-Hilaire
Locations (1):
- Clinique Saint Hilaire, Rouen, France